CLINICAL TRIAL: NCT00335361
Title: The Intra Vas Device (IVD) As A Means of Male Reproductive Sterilization A Single Armed Feasibility Study
Brief Title: Implantable Device for Male Reproductive Sterilization
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shepherd Medical Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G050215; NIH grant # R44HD046318
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Male Sterilization
Keywords: Male Contraceptive Devices; Intra Vas Device (IVD); Male Sterilization; Vasectomy; Intra Vas Deferens Occlusion; Vas Occlusion

INTERVENTIONS:
Device: Intra Vas Device (IVD)

SUMMARY:
The study is to evaluate a device for male reproductive sterilization and determine if this device is successful at blocking the sperm.

Ninety subjects from two centers in the United Stated will be followed closely for 24 months.

If you are someone interested in a vasectomy, you may be eligible to participate in this clinical study.

DETAILED DESCRIPTION:
This feasibility study is intended to collect pertinent clinical information on the use of the Shepherd Medical Intra Vas Device (IVD) necessary to support the design of a future pivotal study. The IVD is intended to occlude the vas deferens and thus accomplish male reproductive sterilization and to offer an additional method to vasectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject desires to undergo a vasectomy.
2. Freely consents to participate in the Study a
3. Agrees to provide a semen sample at regularized periods for at least 30 months.
4. Willing to use a redundant method of contraception until successful occlusion is confirmed.
5. Agrees to provide follow-up information.
6. Willing and able to understand and agree to follow all aspects of the procedures and Study requirements.
7. At least 18 years of age.

Exclusion Criteria:

1. Has a condition permanently or temporarily making participation in the Study inadvisable.
2. Has a condition permanently or temporarily making a vasectomy inadvisable.
3. Has had a previous successful/unsuccessful vasectomy.
4. Has had an allergic reaction to silicone and/or ethylene.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-09; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Successful IVD implantation with vas deferens occlusion at 6 and 24 months post-implant.
The IVD consists of a tubular silicone plug that is inserted into the lumen of the vas deferens to block the flow of semen.
IVD implantation does not require the need to sever or permanently damage the vas deferens like the Ligation/Excision, Clip devices, Cautery
techniques or Fascial Interposition require. One major advantage of the IVD is that it
does not require excision and removal of a portion of the vas. Implantation of the IVD
allows the vas deferens to remain intact and not be permanently damaged.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Douglas G. Stein, MD, PA, Tampa, Florida
  - Regional Urology, LLC, Shreveport, Louisiana
  - Adult and Pediatric Urology, Sartell, Minnesota